CLINICAL TRIAL: NCT06295913
Title: Health Effects of Chronic Supplementation with a Natural Extract High in Hydroxytyrosol in Individuals At High Risk of Developing Age-related Diseases
Brief Title: Hydroxytyrosol Dietary Supplement and Prevention of Age-Related Diseases
Acronym: HT15
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: Genosa I+D (Unknown)
Responsible Party: Principal Investigator, María Raquel Mateos Briz, Investigator, National Research Council, Spain
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: HT15
Record Dates: First submitted 2024-02-20; First posted 2024-03-06 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-02

CONDITIONS: Overweight; PreDiabetes
Keywords: Hydroxytyrosol; Prediabetes; Age-related diseases; Antioxidant
MeSH Terms: conditions — Overweight; Prediabetic State

STUDY DESIGN:
Intervention Model Description: Group 1, hydroxytyrosol-rich extract pill; Group 2, placebo pill
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be randomly allocated to treatment A and B. Both pills will have the same aspect and will be packed similarly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Capsule of an olive extract with a high content of hydroxytytorosol. Group 1 (Experimental): Intake of one capsule/day containing 15 mg of hydroxytyrosol before breakfast for 16 weeks.
  Interventions: Dietary Supplement: Group 1, hydroxytyrosol-rich extract capsule
- Capsule of placebo. Group 2 (Active Comparator): Intake of one capsule placebo/day without hydroxytyrosol before breakfast for 16 weeks.
  Interventions: Dietary Supplement: Group 2, capsule of placebo

INTERVENTIONS:
Dietary Supplement: Group 1, hydroxytyrosol-rich extract capsule — Following a two-week washout period, the subjects will receive a bottle containing capsules (Group 1). Blood, urine, and fecal samples will be collected from each participant during their stay at the Human Nutrition Unit at the beginning and end of the study. Subjects will be instructed to refrain from consuming products rich in hydroxytyrosol (such as virgin olive oil and olives) and to maintain their usual dietary habits throughout the study. Additionally, olive oil (1L/week) will be provided to each volunteer that will consume during intervention study as the sole source of dietary fat, used for cooking, salad dressing, toasts, etc. in order to control the extra consumption of hydroxytyrosol apart from that provided by the capsule.
  Arms: Capsule of an olive extract with a high content of hydroxytytorosol. Group 1
Dietary Supplement: Group 2, capsule of placebo — Following a two-week washout period, the subjects will receive a bottle containing capsules (Placebo) (Group 2). Blood, urine, and fecal samples will be collected from each participant during their stay at the Human Nutrition Unit at the beginning and end of the study. Subjects will be instructed to refrain from consuming products rich in hydroxytyrosol (such as virgin olive oil and olives) and to maintain their usual dietary habits throughout the study. Additionally, olive oil (1L/week) will be provided to each volunteer that will consume during intervention study as the sole source of dietary fat, used for cooking, salad dressing, toasts, etc. in order to control the extra consumption of hydroxytyrosol.
  Arms: Capsule of placebo. Group 2

SUMMARY:
The primary objective of this study is to ascertain the effects of chronic consumption of a hydroxytyrosol-rich extract from olive in a population at high risk of developing age-related pathologies such as type 2 diabetes and cardiovascular diseases. The markers measured will be associated with oxidative stress, inflammation, and homeostasis glucose and lipid profiles. Improvements in these parameters could potentially prevent the onset of pathologies associated with aging.

DETAILED DESCRIPTION:
Fifty subjects 40-75 years old overweight (BMI between 24-29,9 kg/m2) and prediabetes (fasting blood sugar between 100-126 mg/dl and/or glycated hemoglobin between 5,7-6,4%) will be recruited. Detailed inclusion and exclusion criteria are provided below.

Participants will be randomly divided into two groups, one to consume the Hytolive® capsule and the other a placebo. The intervention study has been designed for daily consumption before breakfast of one capsule for 16 weeks. The study includes a two-week washout period during which subjects will not be allowed to consume olives or virgin olive oil.

At the beginning and end of the study, upon arrival at the ICTAN-CSIC Human Nutrition Unit, volunteers will provide a urine sample corresponding to the first morning void, and a nurse will draw a fasting blood sample (20 mL distributed in tubes with various anticoagulants for measurements). Additionally, their blood pressure will be measured, and a complete anthropometric and body composition study will be conducted. Furthermore, volunteers will provide a stool sample from the preceding days (these samples will not be used in this study but will be stored at -80°C for potential future determination of the intestinal microbiota metagenomic profile). Subsequently, dietary controls will be conducted, physical activity and emotional well-being tests will be administered, and fatigue will be evaluated. Additionally, there will be an interim visit aimed at verifying adherence to supplementation. For this purpose, volunteers will provide a urine sample corresponding to the first morning void on an empty stomach, in which levels of hydroxytyrosol and its derivatives will be determined. Likewise, dietary and physical activity controls will be conducted to confirm that volunteers are not altering their habits.

ELIGIBILITY:
Inclusion Criteria:

* Prediabetes (defined as fasting glucose levels according to the American Diabetes Association guideline, with fasting blood glucose ≥100 and <126 mg/dL, or hemoglobin A1c levels ranging from 5.7% to 6.4%)
* Overweight (body mass index BMI 24-29.9 kg/m2)

Exclusion Criteria:

* Any prior diagnosis of diabetes, hypertension, hyperlipidemia, other cardiovascular diseases, thyroid gland disorders, asthma, arthritis, or inflammatory conditions, cirrhosis, or other liver diseases
* Weight loss > 2.5 kg in the last 6 months
* Being on pharmacological treatment of any kind
* Taking dietary supplements containing antioxidants other than vitamins
* Being a smoker or habitual alcohol consumer; being HIV positive
* Being pregnant or breastfeeding
* Blood pressure ≥ 140 mmHg (systolic) and ≥ 90 mmHg (diastolic)
* Total cholesterol ≥ 240 mg/dL, LDL cholesterol ≥ 160 mg/dL, or TG ≥ 200 mg/dl

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
LDL-ox as marker of oxidative status | Up to six months
  Differences between subjects supplemented with hydroxytyrosol and non-supplemented subjects

SECONDARY OUTCOMES:
Mental well-being determined by Warwick-Edinburgh Mental Well-being Scale | Up to two months
  Differences between subjects supplemented with hydroxytyrosol and no-supplemented subjects
Sleep quality determined by Pittsburgh Sleep Quality Index | Up to two months
  Differences between subjects supplemented with hydroxytyrosol and no-supplemented subjects
Fatigue test determined by Borg Rating Of Perceived Exertion | Up to two months
  Differences between subjects supplemented with hydroxytyrosol and no-supplemented subjects
Fasting glucose | Up to six months
  Differences between subjects supplemented with hydroxytyrosol and no-supplemented subjects
Fasting insulin | Up to six months
  Differences between subjects supplemented with hydroxytyrosol and no-supplemented subjects
Glycated hemoglobin (HbA1c) | Up to six months
  Differences between subjects supplemented with hydroxytyrosol and no-supplemented subjects
Glucagon-like peptide-1 (GLP-1) | Up to six months
  Differences between subjects supplemented with hydroxytyrosol and no-supplemented subjects
Total cholesterol | Up to six months
  Differences between subjects supplemented with hydroxytyrosol and no-supplemented subjects
High density lipoproteins (HDL) | Up to six months
  Differences between subjects supplemented with hydrpxytyrosol and no-supplemented subjects
Low density lipoproteins (LDL) | Up to six months
  Differences between subjects supplemented with hydroxytyrosol and no-supplemented subjects
Triglycerides | Up to six months
  Differences between subjects supplemented with hydroxytyrosol and no-supplemented subjects
Apoliporpotein A1 | Up to six months
  Differences between subjects supplemented with hydroxytyrosol and no-supplemented subjects
Apoliporpotein B | Up to six months
  Differences between subjects supplemented with hydroxytyrosol and no-supplemented subjects
Total antioxidant status (TAS) | Up to six months
  Differences between subjects supplemented with hydroxytyrosol and no-supplemented subjects
Total oxidative status (TOS) | Up to six months
  Differences between subjects supplemented with hydroxytyrosol and no-supplemented subjects
Oxides of nitrogen (NOx) | Up to six months
  Differences between subjects supplemented with hydroxytyrosol and no-supplemented subjects
Thiobarbituric acid reactive substances (TBARS) | Up to six months
  Differences between subjects supplemented with hydroxytyrosol and no-supplemented subjects
C reactive protein | Up to six months
  Differences between subjects supplemented with hydroxytyrosol and no-supplemented subjects
Interleukine 6 (IL-6) | Up to six months
  Differences between subjects supplemented with hydroxytyrosol and no-supplemented subjects
Tumor necrosis factor alpha (TNF-α) | Up to six months
  Differences between subjects supplemented with hydroxytyrosoland no-supplemented subjects
Alanine aminotransfesare (transaminases ALT) | Up to six months
  Differences between subjects supplemented with hydroxytyrosol and no-supplemented subjects
Aspartate aminotransferase (transaminase AST) | Up to six months
  Differences between subjects supplemented with hydroxytyrosol and no-supplemented subjects

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Mateos, PhD, Principal Investigator — Institute of Food Science, Technology and Nutrition (ICTAN-CSIC)
Locations (1):
- Institute of Food Science, Technology and Nutrition, National Research Council (ICTAN-CSIC), Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moratilla-Rivera I, Perez-Jimenez J, Ramos S, Portillo MP, Martin MA, Mateos R. Hydroxytyrosol supplementation improves antioxidant and anti-inflammatory status in individuals with overweight and prediabetes: A randomized, double-blind, placebo-controlled parallel trial. Clin Nutr. 2025 Sep;52:17-26. doi: 10.1016/j.clnu.2025.07.006. Epub 2025 Jul 12. PMID 40690822